CLINICAL TRIAL: NCT05189080
Title: Text Message Follow-up for Patients Who Have Missed Well-Child Visits: Open Trial
Brief Title: Twilio Well-Child Visit Pilot Open Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00074978-OT
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-05

CONDITIONS: Child Health; Text Messaging
Keywords: child health; well child visits; text messaging
MeSH Terms: interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: The first phase of the study will be an open trial to assess feasibility and acceptability of three different reminder messages, analyze preliminary data, and collect feedback from participants using interviews to identify the top one or two performing messages. Each reminder message will at minimum direct parents/guardians to reschedule by phone or by the patient portal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Trial (Experimental): Patients within the Wake Forest Baptist Health system who no-showed for scheduled well child visits at Pediatrics-Downtown Health Plaza, Family Medicine-Piedmont Plaza, Pediatrics-Winston East, Family Medicine-Peace Haven, and Pediatrics-Clemmons.
  Interventions: Other: Text message reminders; Other: Interviews; Other: Survey

INTERVENTIONS:
Other: Text message reminders — Text messages will be sent to parents/guardians of children ages 0 to 17 years who no-showed for their well child visits.
Other: Interviews — Interviews will be conducted with a subset of participants to identify the top one or two performing text messages.
Other: Survey — Alongside notification text messages regarding no-showed visits, participants will be invited to participate in a survey about their experience with the health system. This survey will assess reasons for missing the WCV and primary caregiver's perspective on the experience at the prior visit.

SUMMARY:
This project will use Twilio as a platform for a text messaging campaign to implement timely follow up with parents/guardians of children ages 0 to 17 years who have no-showed for WCVs. The first phase of the study will be an open trial to assess feasibility and acceptability of three different reminder messages, analyze preliminary data, and collect feedback from participants using interviews to identify the top one or two performing messages. Each reminder message will at minimum direct parents/guardians to reschedule by phone or by the patient portal. These findings will be used to conduct the second phase of the study, a randomized controlled trial.

DETAILED DESCRIPTION:
Well-Child visits (WCV) are an opportunity to maximize the health and future well-being and development of children. Missed visits, however, can result in negative outcomes for patients and families and for the healthcare system. For patients, missed primary care visits can result in greater Emergency Department (ED) visits and hospitalizations, and in delays in diagnosing a variety of medical conditions, including identification of child abuse and neglect. For healthcare systems, missed visits result in decreased efficiency, lower quality measures, decreased provider productivity, and loss in revenue. Although smart phones are nearly ubiquitous, even among more economically disadvantaged populations, literature to date has reported only on using text messages for pre-visit reminders. There is a tremendous opportunity to study use of text messaging to engage families in follow-up for missed WCV. Even more so, testing the use of text messages with different content is missing, as well as using text messages to invite patients to share reasons for missing the last WCV.

ELIGIBILITY:
Inclusion Criteria:

Patients included in text messaging campaign (caregivers receive text messages):

* Are 0-17 years
* No-showed for a well-child visit scheduled at one of five locations: Pediatrics-Downtown Health Plaza, Family Medicine-Piedmont Plaza, Pediatrics-Winston East, Family Medicine-Peace Haven, or Pediatrics-Clemmons
* Have a phone number on record for a primary caregiver
* With primary language for contact that is English or Spanish

Caregivers must be 18 years or older

Exclusion Criteria:

Patients who:

* Are 18+ years old
* No-showed for a different type of visit, or no-showed for a WCV at a different practice location
* Already rescheduled their appointment by the time the sample list was generated
* Have primary language specified that is not English or Spanish.

Caregivers who are under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Number of rescheduled well child visits | 6 weeks after no-showed well child visit
  If parent/guardian rescheduled well child visit
Number of completed (rescheduled) well child visits | 6 weeks after no-showed well child visit
  If parent/guardian completed (rescheduled) well child visit

SECONDARY OUTCOMES:
Number of child patient emergency department visits | 6 weeks after no-showed well child visit
  If child patient had an emergency department visit
Number of child patient hospitalizations | 6 weeks after no-showed well child visit
  If child patient required hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Poehling, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT05189080/ICF_000.pdf